CLINICAL TRIAL: NCT02390765
Title: Children's Growth and Behavior Study
Brief Title: Children s Growth and Behavior Study
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150096; 15-CH-0096
Record Dates: First submitted 2015-03-17; First posted 2015-03-18 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Obesity; Eating Behaviors; Healthy Volunteers
Keywords: Stress Response; Binge Eating; Eating Behavior; Obesity; Disordered Eating; Natural History
MeSH Terms: conditions — Obesity; Feeding Behavior; Fractures, Stress; Bulimia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All pediatric participants: All pediatric participants in the study will be evaluated as one group
- Parents of participants: Parents provide information about their children and supply DNA / blood samples for future analyses

SUMMARY:
Background:

- Studies show that many factors affect children's eating behavior and health. These include sleep, mood, thinking skills, and genetics. Studying children over time may identify children at higher risk for eating-related health concerns.

Objective:

- To understand how genes and environment influence eating behavior and health over time.

Eligibility:

- Children ages 8-17 in good general health.

Design:

* Screening visit 1: Medical history, physical exam, body measurements, and questions.
* 14 days: Participants will wear a wrist monitor and answer smartphone prompts about eating and mood. They may give a stool sample.
* Screening visit 2:
* Body measurements.
* Saliva, urine, and blood samples.
* Heart tests.
* Meals provided (after fasting overnight).
* Questionnaires and interview.
* Behavior, thinking, and exercise tests.
* X-ray of left wrist and full body.<TAB>
* Some parents may have medical history, physical exam, and questions at screening visits. They may answer questions at the yearly visits.
* Participants will have up to 6 yearly visits. They will give a urine sample and body measurements, and repeat the X-rays. They will have questions and behavior and thinking tasks. They may give stool samples. Visits will range from 3 to 8 hours.
* Participants may choose to participate in other studies:
* Stress and Hormones, 1 visit: While resting, participants will give saliva samples and have their heart monitored. Then they will do math. They will repeat the resting part, then do a computer task.
* Brain Imaging, 2 visits: Twice, participants will perform tasks with a magnetic cone on their head then answer questions. Once, they will have an MRI, lying still in a scanner with a coil on their head. Before the first visit, participants will collect at-home saliva samples once a day for three days. During both visits, participants will perform tasks and answer questions that gauge their thinking skills and mood.
* Experiment 3 (sleep/fatigue): Participants will complete 2 additional visits. During these visits, participants will complete a task on the computer for 2 hours, or watch a movie for two hours. After completion of the task/movie, they will answer questions and be provided with food.

Participants will be compensated for the time and inconvenience involved with completing study procedures.

DETAILED DESCRIPTION:
This study aims to disentangle the varying disinhibited eating patterns, or eating behavior endophenotypes, that lead to excessive weight gain and obesity-related comorbidities in youth. Extensive baseline evaluations, including three separate experimental paradigms, and annual follow-up assessments will assist with identifying biopsychosocial mechanisms that appear to increase risk for, and maintain, these eating behaviors and lead to weight gain. Illumination of early risk factors for specific eating behavior endophenotypes and their associated health outcomes will inform the development of targeted interventions for pediatric obesity. Participants for the current study will include 500 healthy obese and non-obese boys and girls (8 to 17yo at baseline) and their parents/caregivers. Youth will first complete two visits in order to ensure study eligibility and to evaluate self-regulatory, motivational, and neurocognitive factors that appear to be salient to the development and maintenance of disinhibited eating behavior, including: psychological distress, sleep behavior, food reinforcement, reward sensitivity, executive functioning, attention bias, and a range of related genetic and physiological factors. Eating behavior will be observed in the laboratory using several validated paradigms. For two weeks, participants will monitor their sleep using wrist actigraphy, as well as record their mood, eating behavior, and eating cognitions using smart phones (via ecological momentary assessment methods). Youth will then be invited to complete up to three separate experimental paradigms designed to further elucidate cognitive, emotional, and physiological processes associated with disinhibited eating behavior. All participants will then complete annual evaluations of weight and adiposity for a total of six years, with more extensive evaluations of self-regulatory, motivational and neurocognitive functioning every three years. Studying children and adolescents longitudinally will allow for examination of the independent and shared risk factors for pediatric disinhibited eating and excess weight. Data from these evaluations will not only be used to test specific hypotheses, but will also be hypothesis-generating in that they will inform the development of additional empirical questions and subsequent experiments. Thus, the current protocol will offer the flexibility to examine potentially critical contributions to weight gain in children as they continue their biopsychosocial development.

ELIGIBILITY:
* Eligibility Criteria for Parents/Guardians of Child Participants:

INCLUSION CRITERIA:

Parents/Guardians will qualify if they meet the following criteria.

1. Age >=18 years
2. Have a child enrolled in this protocol (15-CH-0096).

EXCLUSION CRITERIA:

Parents/Guardians will be excluded for the following reasons:

1. If their child is not eligible to participate in the study (see below)
2. If they are believed by the medical study team to have a medical or psychiatric problem that will not allow them to complete study procedures safely (these will be determined on a case-by-case basis)

   Eligibility Criteria for Child Participants:

   INCLUSION CRITERIA:

   Volunteers will qualify if they meet the following criteria.
   * Age 8-17 years (NB: children may continue to participate as adults during follow-up).
   * Weight, height and BMI >= 5th percentile for age and sex according to Centers for Disease Control and Prevention 2000 US standards.
   * Cognitively capable of completing study procedures (FSIQ >= 70).
   * Good general health based on a normal history and physical examination (with the exception of overweight and minor, well-controlled illnesses).

   EXCLUSION CRITERIA:

   Individuals will be excluded (and provided treatment referrals as needed) for the following reasons:
   * History of major cardiovascular disease or any other serious obesity-related complication as assessed during history and physical exam. Individuals with untreated or major illnesses relating to the endocrine and/or cardiovascular systems are excluded because these illnesses will likely influence outcomes. Such obesity-related comorbidities include hypertension (defined by age- sex- and height- specific standards; and fasting hyperglycemia consistent with diabetes (fasting glucose > 126 mg/dL).
   * Presence of other major illnesses: renal, hepatic, gastrointestinal, most endocrinologic (e.g., Cushing syndrome, untreated hyper- or hypothyroidism), hematological problems or pulmonary disorders (other than asthma not requiring continuous medication). Non-serious medical illnesses, such as seasonal allergies, will be reviewed on a case-by-case basis.
   * Regular use of any medication known to affect body weight or eating behavior (e.g., many medications prescribed for attention deficit hyperactivity disorder, or ADHD). Medication use for non-serious conditions (e.g., acne) will be considered on a case-by-case basis.
   * Current pregnancy or a history of pregnancy. A negative pregnancy test before starting the study will be required for postmenarcheal girls.
   * Current and regular use of tobacco products and/or alcohol.
   * A significant reduction in weight during the past three months, for any reason, exceeding 5% of body weight.
   * A history of significant or recent brain injury that may considerably influence performance on neurocognitive measures (i.e., any history of loss of consciousness >=30 minutes associated with a head injury, any history of memory loss or hospitalization associated with a head injury, or >=2 concussions within last year).
   * Presence of any significant, full-threshold psychiatric disorder based on DSM criteria such as schizophrenia, bipolar disorder, alcohol or substance abuse, anorexia or bulimia nervosa, or any disorder that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study. These individuals will not be permitted to enroll in the current study and will be referred for treatment. Individuals who present with other psychiatric disorders, including sub-threshold psychiatric disorders, will be permitted to enroll in the study. Sub-threshold psychiatric disorders include symptoms that do not meet diagnostic threshold based on the DSM criteria for mental disorders, but which are nevertheless significantly impairing or distressing. If, based on the opinion of the investigators, a participant requires treatment for his/her psychiatric symptoms, the individual will be referred for treatment. Participants who develop any psychiatric disorder or significant psychiatric symptoms at any follow-up assessment during the study will not be excluded, but will be provided with treatment referrals.
   * Any other condition in the child or parents/guardians that, in the opinion of the investigators, would impede compliance or possibly hinder completion of the study (e.g., significant Learning Disorder).

   Additional exclusions for (optional) stool sample collection include:

   Stool Sample only:
   * Diagnosis or history of inflammatory bowel disease, including ulcerative colitis or Crohn's disease, celiac sprue, irritable bowel syndrome, or other inflammatory disorders of the intestine.
   * Diarrhea within 1 week prior to sampling.
   * Antibiotic use within 4 weeks prior to sampling.

   In addition, Experiments 1 and 2 have specific additional exclusions:

   Experiment 1 only:
   * Regular use of medications that could influence autonomic or endocrine functioning, including alpha and beta blockers, oral contraceptives, or prescription pain medication.
   * Scoring as "highly active" on the International Physical Activity Questionnaire (due to decreased cortisol reactivity).

   Experiment 2 only:
   * Participants will be excluded if MRI and MEG is contraindicated (metal in/on body, braces, presence of non-organic [e.g., cochlear] implants or cerebral clips, permanent tattooed makeup or general tattoos that are recent and/or in a dangerous location on the body or made with colors whose content in iron cannot be definitely ruled out.
   * Youth will be excluded if they are left-handed.

   All participants will receive a written explanation of the purposes, procedures, and potential hazards of the study. Communication of this information and of the participant's assent as well as the consent of the parent or guardian will be documented in the medical record and copies of all signed documents given to each family. All participants will be informed of their right to withdraw from the study.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-04-21 (Actual); Primary Completion 2030-12-12 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in eating behavior of pediatric participants | up to 6 years of follow-up
  Multiple outcome measures

SECONDARY OUTCOMES:
Experiment 2 (Hormone and Brain Development Study): oscillatory power activity in hypothesized brain regions-of-interest and food intake in the laboratory | During palatable (vs non-palatable) food cues attention bias paradigm
  Explore whether gonadal hormone concentrations moderate the association between activation in ROIs and LOC-eating in the laboratory. Hyp 3a: The associations among activation in ROIs and LOC-eating severity will be stronger among girls with higher concentrations of estradiol. Hyp 3a: The associations among activation in ROIs and total energy intake will be stronger among girls with higher concentrations of estradiol. Hyp 3c: The associations among activation in ROIs and LOC-eating severity will be stronger among boys with lower concentrations of testosterone. Hyp 3d: The associations among activation in ROIs and total energy intake will be stronger among boys with lower concentrations of testosterone.
Experiment 2 (Hormone and Brain Development Study): oscillatory power activity in hypothesized brain regions-of-interest and food intake in the laboratory | During palatable (vs non-palatable) food cues attention bias paradigm
  Investigate if model-based decision making mediates the link between activation in ROIs while attending to images of food and LOC-eating in the laboratory. Hyp 2a: Model-based decision making (DM) will mediate the association between activation in all ROIs and severity of LOC-eating. Hyp 2a: Model-based DM will mediate the association between activation in all ROIs and total energy intake.
Experiment 2 (Hormone and Brain Development Study): oscillatory power activity in hypothesized brain regions-of-interest | During palatable (vs non-palatable) food cues attention bias paradigm
  Examine if activation in neural regions of interest (ROIs; striatum, prefrontal cortex, and hippocampus) while attending to food images is linked to decision making (DM) during a decision-making task. Hyp 1a: Striatum activation will be related to model-free learning. Hyp 1b: Activation in all ROIs will be linked to model-based learning.
Experiment 2 (Hormone and Brain Development Study): oscillatory power activity in hypothesized brain regions-of-interest | During palatable (vs non-palatable) food cues attention bias paradigm
  Differences in neural activity in youth with- and without Loss of Control Eating. In the model examining the initial attention capture period of the palatable food attention bias paradigm, condition will be coded as high-palatable food, low-palatable food, and neutral non-food trials. In the model examining the sustained attention deployment period of the palatable food attention bias paradigm, the conditions will be coded as high palatable-congruent and -incongruent trials, as well as low palatable-congruent and -incongruent trials.
Experiment 2 (Hormone and Brain Development Study): oscillatory power activity in hypothesized brain regions-of-interest | During social threat attention bias paradigm
  Differences in neural activity in youth with- and without Loss of Control Eating. In the model examining the initial attention capture period, condition will be coded as angry, happy, and neutral trials. In the model examining the sustained attention deployment period, the conditions will be coded as angry-congruent and -incongruent trials, as well as happy-congruent and -incongruent trials.
Experiment 3 (Sleep/fatigue): fatigue and task resistance | Immediately before and after completion of the computer task and movie (approximately 2hours)
  Difference in self-report of fatigue and resistance during the computer task and movie. According to a prior power calculations, the sample size (40 participants) was expected to have 80% power to detect a significant difference between the cognitive fatigue and non-fatigue conditions based on effect sizes from previous studies of adults (Cohen s d=0.8-2.5) [Faber, Maurits, & Lorist, 2012; Van der Linden & Eling, 2006].Faber LG, Maurits NM, Lorist MM. Mental fatigue affects visual selective attention. PLoS One 2012;7:e48073. doi: 10.1371/journal.pone.0048073Van der Linden D, Eling P. Mental fatigue disturbs local processing more than global processing. Psychol Res 2006;70:395-402.
Experiment 3 (Sleep/fatigue): behavioral performance | During the computer task (~2hours).
  Reaction time and proportion of correct responses during the fatigue task.
Experiment 3 (Sleep/fatigue): energy intake. | Immediately following completion of the computer task and movie.
  Difference in total energy intake (kcals) during the laboratory meals following the computer task and movie.A priori power computations were based on the effect size from a previous laboratory study evaluating energy intake differences between adults randomized to a high or low cognitive reduction condition [Ward and Mann, 2000]. To detect a difference in energy intake, using a randomized crossover design with power of 0.9 and a 2-sided significance level of =.05, 88 participants were required.Ward A, Mann T. Don't mind if i do: Disinhibited eating under cognitive load. J Pers Soc Psychol 2000;78:753-63. doi: 10.1037//0022-3514.78.4.753

CONTACTS AND LOCATIONS:
Overall Officials: Bobby K Cheon, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data sets that underlie results in a publication are to be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: NIH subject data will become available starting 6 months after publication of a results paper and will be available from the NIH site for 2 years.
Access Criteria: NIH data with personal identifiers removed will be shared upon reasonable request to the PI, who will review requests. A data sharing agreement will be required to be negotiated with NICHD before sharing takes place.

REFERENCES:
- [Background] Tanofsky-Kraff M, Yanovski SZ, Wilfley DE, Marmarosh C, Morgan CM, Yanovski JA. Eating-disordered behaviors, body fat, and psychopathology in overweight and normal-weight children. J Consult Clin Psychol. 2004 Feb;72(1):53-61. doi: 10.1037/0022-006X.72.1.53. PMID 14756614
- [Background] Tanofsky-Kraff M, Shomaker LB, Olsen C, Roza CA, Wolkoff LE, Columbo KM, Raciti G, Zocca JM, Wilfley DE, Yanovski SZ, Yanovski JA. A prospective study of pediatric loss of control eating and psychological outcomes. J Abnorm Psychol. 2011 Feb;120(1):108-18. doi: 10.1037/a0021406. PMID 21114355
- [Background] Tanofsky-Kraff M, Cohen ML, Yanovski SZ, Cox C, Theim KR, Keil M, Reynolds JC, Yanovski JA. A prospective study of psychological predictors of body fat gain among children at high risk for adult obesity. Pediatrics. 2006 Apr;117(4):1203-9. doi: 10.1542/peds.2005-1329. PMID 16585316
- [Derived] Parker MN, Tanofsky-Kraff M, Bloomer BF, Te-Vazquez J, Adekola PE, Nwosu EE, Lazareva J, Jones JL, Moore A, Schvey NA, Brady SM, Yang SB, Turner SA, Yanovski JA, Kelly NR. The Effect of Experimentally Induced Cognitive Fatigue on Energy Intake Among Youth With and Without Recent Reported Dietary Restraint. Int J Eat Disord. 2025 Oct;58(10):2003-2008. doi: 10.1002/eat.24508. Epub 2025 Jul 16. PMID 40878932
- [Derived] Parker MN, Kelly NR, Moore A, Loch LK, Vazquez JT, Bloomer BF, Nwosu EE, Lazareva J, Yang SB, Courville AB, Moursi NA, Brady SM, Olsen CH, Shank LM, Tanofsky-Kraff M, Yanovski JA. Cognitive fatigue did not significantly influence youth's total energy intake or snack food consumption during a randomized trial. J Behav Med. 2025 Aug;48(4):683-693. doi: 10.1007/s10865-025-00577-8. Epub 2025 Jun 9. PMID 40489009
- [Derived] Smith MR, Bittner JMP, Loch LK, Haynes HE, Bloomer BF, Te-Vazquez J, Bowling AI, Brady SM, Tanofsky-Kraff M, Chen KY, Yanovski JA, Cheon BK. Independent and Interactive Associations of Subjective and Objective Socioeconomic Status With Body Composition and Parent-Reported Hyperphagia Among Children. Child Obes. 2024 Sep;20(6):394-402. doi: 10.1089/chi.2023.0086. Epub 2023 Nov 9. PMID 37943608
- [Derived] Rubin AG, Schvey NA, Shank LM, Altman DR, Swanson TN, Ramirez E, Moore NA, Jaramillo M, Ramirez S, Davis EK, Broadney MM, LeMay-Russell S, Byrne ME, Parker MK, Brady SM, Kelly NR, Tanofsky-Kraff M, Yanovski JA. Associations between weight-based teasing and disordered eating behaviors among youth. Eat Behav. 2021 Apr;41:101504. doi: 10.1016/j.eatbeh.2021.101504. Epub 2021 Mar 29. PMID 33831812
- [Derived] Schvey NA, Shank LM, Tanofsky-Kraff M, Ramirez S, Altman DR, Swanson T, Rubin AG, Kelly NR, LeMay-Russell S, Byrne ME, Parker MN, Broadney MM, Brady SM, Yanovski SZ, Yanovski JA. Weight-based teasing in youth: Associations with metabolic and inflammatory markers. Pediatr Obes. 2021 Mar;16(3):e12729. doi: 10.1111/ijpo.12729. Epub 2020 Oct 15. PMID 33059389
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-CH-0096.html